CLINICAL TRIAL: NCT06602154
Title: Comparison of Bond Failure with Resin-modified Glass Ionomer Cement and Visible Light-cure Composite Bonding Material in Adult Orthodontic Patients - a Split-Mouth, Randomized Controlled Trial
Acronym: RMGIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Rashna Hoshang Sukhia, Associate Professor, Program Director, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-5282-23281; Dr. Aleem Saeed Qureshi (Other: AKUH)
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Orthodontics; Bracket Bonding; Malocclusion; Displaced or Missing Teeth
Keywords: Resin-modified glass ionomer cement; Light cure composite; bracket bonding
MeSH Terms: conditions — Malocclusion; Anodontia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Control group ( light cure composite ) (Active Comparator): Product: Denturum Light Cure Band Adhesive (Ortho Organizers). Composition: 4 mg composite adhesive paste and 6 ml Transbond primer. Storage: Stored at room temperature and protected from humidity.
  Usage: Steps for light -cure composite bonding are:
  1. Prepare teeth with oil-free pumice, and rinse thoroughly for 15 seconds with water.
  2. Air dry tooth surface for 5 seconds until dry field is maintained and isolate with cotton rolls.
  3. Etch enamel surface with 37% phosphoric acid for 15 seconds.
  4. Rinse the etched surface for 20 seconds to remove the acid and precipitates that might have formed during the etching procedure.
  5. Thoroughly dry etched surface with moisture free air. Tooth surface should appear frosty white, if not than reetch for 5 seconds.
  6. Brush thin uniform amount of primer on every tooth surface.
  7. Apply a small amount of adhesive paste onto bracket base and position the bracket on tooth surface.
  8. After accurately placing bracket on tooth surfac
  Interventions: Other: Resin modified glass ionomer

INTERVENTIONS:
Other: Resin modified glass ionomer — The product will be stored by investigators at room temperature in lock and key.
  Product: Riva light cure RMGIC (HV) Composition: 18 mg orthodontic bonding paste and 6 ml enamel bond resin. Storage: Stored at room temperature and protected from humidity.
  Usage: Steps for Resin-modified glass ionomer cement composite bonding:
  1. Prepare all teeth with oil-free pumice, and rinse thoroughly for 15 seconds with water.
  2. Wash thoroughly.
  3. Etch enamel surface with 37% phosphoric acid for 15 seconds.
  4. Rinse the etched surface for 20 seconds to remove the acid and precipitates that might have formed during the etching procedure.
  5. Activate the capsule and immediately mix in an amalgamator. Do not click with applicator before you mix.
  6. Immediately place into capsule applicator and click trigger until paste is seen through the nozzle
  7. Light cure each increment for 20 seconds.

SUMMARY:
In this split mouth study design, 34 orthodontic patients coming for fixed appliance treatment will be bonded with standard light-cure composite bonding material and intervention of Resin Modified Glass Ionomer Cement (RMGIC). Contralateral quadrants will be allocated randomly for either RMGIC or visible light-cure composite bonding in both upper and lower jaw.

Quadrant 1: Randomly selected, contralateral upper and lower quadrants from central incisor to second premolar will be bonded with RMGIC bonding system.

Quadrant 2: Randomly selected, contralateral quadrants from central incisor to second premolar will be bonded with visible light-cure composite bonding material.

Allocation of diagonally opposite quadrants by either bonding system will be assigned randomly. Quadrants to be bonded with Resin-modified glass ionomer cement and light-cure composite bonding material will be switched from patient to patient to ensure randomization. This study is single blinded. The study investigators will not be blinded while the patient will be kept blinded.

On the first visit, a specially designed consent form will be signed by the participant.

Patient interaction for the purpose of study will only be for 1 hour duration while bonding of brackets. After six months amount and location of bond breakages will be evaluated from orthodontic record files.

This study will help us evaluate bond strength of RMGIC as compared to light cure composite. RMGIC can also be considered as the choice of material for bonding in high risk caries patients.

DETAILED DESCRIPTION:
MATERIAL & METHODS:

Study Design: Experimental study (Randomized Control Trial) Settings: Dental clinics, The Aga Khan University Hospital, Karachi (AKUH) Duration of Study: Patients will be recruited in this study for one and half hour. Chart analysis of these patients will then be done after six months of recruitment.

Sample Size:

Sample size was calculated with OpenEpi (version 3.01) sample size calculator using findings of Hegarty and Macfarlane14 who reported a bond failure percentage of 30% with light-cure adhesive and risk ratio of 2.6 (1.7, 3.9) for RMGIC as compared to resin based light cured composite. Keeping the above risk ratio at level of significance (α) 5% and power of study (1-β) 80%, at least 34 subjects were required for our study. The sample size will be inflated by 10% to account for sample attrition; therefore, a total of 37 subjects will be included in the study.

Sampling Technique: Non-probability consecutive sampling

Sample Selection:

Inclusion Criteria:

* Patients aged between 18-35 years
* Patients with fair to good oral hygiene who have no significant sign of gingivitis
* Healthy patients with no co-morbids such as rheumatic fever, blood dyscrasias, congenital heart disease, or diabetes mellitus
* Patients with class I, II and III malocclusions
* All patients who will sign the consent form

Exclusion Criteria:

* Enamel surface defects
* Pregnant patients or lactating mothers
* Syndromic patients
* Subjects with previous history of orthodontic or functional appliance treatment

DATA COLLECTION PROCEDURE:

Data will be collected by well-organized proforma. (Annexure H) Ethical approval will be taken from the institutional Ethical Review Committee (ERC) before commencement of the study. All those patients who sign an informed consent form (Annexure I) will receive detailed information regarding the study.

Due to ethical considerations, only patients requiring fixed appliance orthodontic treatment will be recruited. In this split mouth study design, contralateral quadrants will be allocated randomly for either Resin-modified glass ionomer cement or visible light-cure composite bonding in both upper and lower jaw. Randomization as per annerxure J Quadrant 1: Randomly selected, contralateral upper and lower quadrants from central incisor to second premolar will be bonded with RMGIC bonding system.

Quadrant 2: Randomly selected, contralateral quadrants from central incisor to second premolar will be bonded with visible light-cure composite.

On the first visit, a specially designed consent form will be signed by the participant. The investigator will unseal the envelope from Clinical Trials Unit (CTU), containing information regarding the participants based on randomization.

Ethical considerations:

Study will be carried out as per guidelines of World Medical Association's Declaration of Helsinki and principles of GCP (Good Clinical Practice). Any modifications in the protocol will be re-submitted to the ERC. The trial will be conducted in compliance with regulations and a copy of the final study protocol will be submitted to ERC.

Consent:

After assessment of eligibility criteria, participants will be included in this study after signing consent form. Consent form will be explained to patient in a separate dental room by investigators to ensure privacy. If patient will be unable to decide then consent form will be given to patient and asked to reply after decision in 7 days. One copy of consent will be given to patient after signing and one copy will be kept with the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 12-35 years
* Patients with fair to good oral hygiene who have no significant sign of gingivitis
* Healthy patients with no co-morbids such as rheumatic fever, blood dyscrasias, congenital heart disease, or diabetes mellitus
* Patients with class I, II and III malocclusions

Exclusion Criteria:

* Enamel surface defects
* Pregnant patients or lactating mothers
* Syndromic patients
* Subjects with previous history of orthodontic

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Bracket bond failure | Three months
  The objective of this study is to compare rate of bond failures with Resin-modified glass ionomer cement and visible light-cure bonding.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Aga Khan University Hospital, Karachi, Sindh
  - Aga Khan University Hospital, Karachi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qabool H, Qabool J, Sukhia RH, Fida M. Comparison of bond failure with resin-modified glass ionomer cement and visible light-cured composite bonding systems in orthodontic patients: A split-mouth randomized controlled trial. Dent Med Probl. 2024 Sep-Oct;61(5):651-657. doi: 10.17219/dmp/162970. PMID 39364623